CLINICAL TRIAL: NCT07149376
Title: Clinical Investigation to Assess the Efficacy of a Toothpaste Containing 8% Arginine as Compared to Colgate Cavity Protection Toothpaste in the Reduction of Dentinal Hypersensitivity.
Brief Title: To Assess the Efficacy of a Toothpaste Containing 8% Arginine as Compared to Colgate Cavity Protection Toothpaste in the Reduction of Dentinal Hypersensitivity.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2025-05-SEN-TOMS-CA-DR
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-08

CONDITIONS: Sensitivity, Tooth
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test 1 toothpaste (Active Comparator): During this clinical study, you will be assigned to one of the two study groups. You will be provided with a toothpaste and toothbrush for at home use. You will be instructed to brush your teeth twice daily for one (1) minute each time. You are to repeat the same procedures for the duration of the study.
  Interventions: Device: TOMs of Maine Sensitive SLS Free Xtra Fresh
- Test 2 toothpaste (Active Comparator): During this clinical study, you will be assigned to one of the two study groups. You will be provided with a toothpaste and toothbrush for at home use. You will be instructed to brush your teeth twice daily for two (2) minute each time. You are to repeat the same procedures for the duration of the study.
  Interventions: Drug: Colgate Cavity protection toothpaste

INTERVENTIONS:
Device: TOMs of Maine Sensitive SLS Free Xtra Fresh — Cover the entire length of bristled head with toothpaste. Brush your teeth twice daily (morning and evening) for one (1) minute each time.
  For investigational use only by the study participant. Not for Sale.
  Arms: Test 1 toothpaste
Drug: Colgate Cavity protection toothpaste — Cover the entire length of bristled head with toothpaste. Brush your teeth twice daily (morning and evening) for (2) two minutes each time.
  For investigational use only by the study participant.
  Arms: Test 2 toothpaste

SUMMARY:
The objective of this clinical investigation is to assess the efficacy of a toothpaste containing 8% arginine (Colgate-Palmolive Company, New York, NY, USA) as compared to a commercially available non-desensitizing toothpaste (Colgate Cavity Protection Toothpaste, Colgate-Palmolive Company, New York, NY, USA) in the reduction of dentinal hypersensitivity over an eight (8) week period.

ELIGIBILITY:
Inclusion Criteria:

* Sign an Informed Consent Form;
* Male or female 18 to 70 years of age, inclusive;
* Be in good general health as determined by the study investigators;
* Available for the eight (8) weeks duration of the study;
* Must present two (2) sensitive teeth which must meet ALL of the following criteria:
* Be anterior to the molars and demonstrating dentin exposure due to cervical erosion/abrasion and/or gingival recession;
* Have a qualifying dentin hypersensitivity response to tactile stimuli applied to the cervical surface (gingivo-facial 1/3) as defined by a response score between 10-50grams of force (Yeaple Probe, XiniX Research Inc. Portsmouth, NH, USA);
* Have a qualifying dentin hypersensitivity response to air blast stimuli applied for one second to the cervical surface (gingivo-facial 1/3) as defined by a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale.

Exclusion Criteria:

* Gross oral pathology, chronic disease, and/or history of allergies to any of the test products
* Use of a desensitizing oral care product and/or recipient of any dental desensitizing treatment within the past three months prior to start of the study;
* Advanced periodontal disease and/or treatment for periodontal disease (including surgery) within the past twelve months
* Sensitive teeth with a mobility greater than one Teeth with extensive/defective restorations (including prosthetic crowns), suspected pulpitis, caries, cracked enamel, or used as abutments for removable partial dentures;
* Current use of anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti- inflammatory drugs, or daily use of analgesics
* Participation in any other oral clinical study for the duration of this study
* Self-reported pregnancy and/or currently breastfeeding;
* Allergies to oral care products, personal care consumer products, and/or their ingredients
* Medical condition which prohibits not eating/drinking for 4 hours

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Tactile stimulation by the Yeaple Probe | baseline, 3 day, 4 weeks, 8 weeks
  Hypersensitivity defined by a response score in the range of 10-50 grams of force.
Air blast stimulation | baseline, 3 day, 4 weeks, 8 weeks
  Jet of air delivered by a standard dental unit syringe at a measured temperature of 19-21°C (70°F [± 3°F]) [hypersensitivity defined by a response score of 2 or 3 on the Schiff Cold Air Sensitivity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Farid Ayad, Principal Investigator — FAR ORAL SYSTEMIC HEALTH CONSULTING INC.
Locations (1):
- FAR Oral and Systemic Health Consulting, Inc, Costa Mesa, California, United States